CLINICAL TRIAL: NCT04391803
Title: EvaLuate EndoVascular Treatment of Acutely Ruptured Shallow Intradural Aneurysms With the Pipeline™ Flex Embolization Device With Shield TEchnology™ (ELEVATE)
Acronym: ELEVATE
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Sponsor-initiated suspension to halt enrollment. Subjects that were enrolled were followed to completion. Last Subject Last Visit occurred on 20-Oct-2025.
Sponsor: Medtronic Neurovascular Clinical Affairs (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MDT19025TRACER
Record Dates: First submitted 2020-04-21; First posted 2020-05-18 (Actual); Last update posted 2026-01-27 (Actual); Status verified 2026-01

CONDITIONS: Intracranial Aneurysm; Ruptured Aneurysm
Keywords: wide neck; intradural aneurysm
MeSH Terms: conditions — Intracranial Aneurysm; Aneurysm, Ruptured

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (1):
- Pipeline™ Flex Embolization Device with Shield Technology™ (Experimental): This is a prospective, single-arm study in which subjects have consented and deployment of the Pipeline™ Flex Embolization Device with Shield Technology™ is attempted.
  Interventions: Device: Pipeline™ Flex Embolization Device with Shield Technology™

INTERVENTIONS:
Device: Pipeline™ Flex Embolization Device with Shield Technology™ — The Pipeline™ Flex Embolization Device with Shield Technology™ is intended for endovascular treatment of adults with intracranial acutely ruptured aneurysms not amenable to clipping and coiling.
  Other Names: Pipeline™ Shield Device

SUMMARY:
The purpose of the study is to assess the safety and effectiveness of the Pipeline™ Flex Embolization Device with Shield Technology™ in the treatment with acutely ruptured intracranial aneurysms.

DETAILED DESCRIPTION:
The ELEVATE study is a prospective, multi-center, single-arm trial of the Pipeline™ Shield Device for the treatment of adults with acutely ruptured intracranial aneurysms. The primary objective of the ELEVATE study is to assess the safety and effectiveness of treatment with the Pipeline™ Shield Device of acutely ruptured intracranial aneurysms that are not amenable for clipping and coiling.

ELIGIBILITY:
Inclusion Criteria:

1. Subject has a previously untreated, wide neck, side-wall, intradural aneurysm that is deemed unfavorable for both surgical clipping and endovascular coiling, as confirmed on DSA.
2. Subject has a ruptured intracranial aneurysm with vessel diameter suitable for treatment with the study device.
3. Subject is ≥ 22 and ≤ 80 years of age.
4. Subject has an acutely ruptured aneurysm with Hunt and Hess Scale 1, 2 or 3.
5. Subject or subject's Legally Authorized Representative (LAR) has provided written informed consent.

Exclusion Criteria:

1. Subject's vessel characteristics preclude safe endovascular access to the aneurysm to treat with the Pipeline™ Shield Device.
2. Subject has aneurysm vessel characteristics that would preclude the device from fully conforming to the parent vessel to reduce any risk of embolic complications, retreatment, or device movement.
3. Subject has true bifurcation or aneurysms with vessels that cannot be separated from the fundus with placement of the study device.
4. Subject with intraparenchymal hemorrhage.
5. Subject is unable to undergo nasogastric/orogastric tube placement prior to device placement.
6. Subject has a pre-morbid mRS >2.
7. Subject requires treatment of another aneurysm (with another treatment modality) within the affected territory of the target aneurysm.
8. Subject has a target ruptured aneurysm that is thought to be mycotic, including those caused by left atrial myxoma, or subject has an active systemic bacterial infection.
9. Subject with a requirement for continuous anti-coagulation.
10. Subject has a malignant brain tumor or vascular malformation (e.g. arteriovenous malformation).
11. Subject's target ruptured aneurysm has not been determined by the treating physician to be the source of SAH.
12. Subject with known allergy to platinum or cobalt chromium alloy (including the major elements platinum, cobalt, chromium, nickel or molybdenum).
13. Subject has a known hypersensitivity to ticagrelor or aspirin.
14. Subject is unable to undergo DSA or DSA is determined unsuitable by the treating physician.
15. Subject has a serious or life-threatening comorbidity that could confound study results.
16. Subject is at high risk of noncompliance per treating physician due to reasons including but not limited to a history of substance abuse.
17. Subject is unable to complete scheduled follow-up assessments due to comorbidities, geographical limitations, or a life expectancy of less than 24 months.
18. Subject is pregnant, or breastfeeding at the time of admission or plans to become pregnant during their participation in the study.
19. Subject is participating in another clinical study at the time of enrollment.
20. Presumed septic embolus, or suspicion of microbial superinfection.
21. Subject with a known COVID-19 viral infection, confirmed by testing.
22. Subject in whom a pre-existing stent is in place in the parent artery at target aneurysm location.

Ages: 22 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2022-05-06 (Actual); Primary Completion 2025-10-20 (Actual); Study Completion 2025-10-20 (Actual)

PRIMARY OUTCOMES:
Incidence of complete angiographic occlusion without significant stenosis, and no rebleeding or retreatment of the target aneurysm | at 365-day
  Occlusion is measured by the Raymond Roy Scale. Significant stenosis is classified as ≤ 50%.
Incidence of neurological death or disabling stroke post-procedure. | at 365-day
  Disabling stroke is defined as any post-procedural ischemic or hemorrhagic event that results in poor functional outcome (i.e. mRS ≥ 3 points) assessed at 90 days post stroke event.

SECONDARY OUTCOMES:
Pipeline™ Flex Device Deployment Success Rate | Day 0 During Procedure
Incidence of rebleed of target aneurysm | through 180-day and 365-day post procedure
Incidence of neurological hemorrhagic serious adverse events | through 180-day and 365-day post procedure
Incidence of ipsilateral major stroke or neurological death post-procedure after 30 days | through 180-day and 365-day post procedure
Incidence of any ipsilateral stroke post-procedure after 30 days | through 180-day and 365-day post procedure
Good clinical outcome (modified Rankin Scale (mRS) 0-2) | at 30-day, 180-day and 365-day post procedure
  Scale for measuring general neurologic function:
  0- No symptoms at all
  1. No significant disability despite symptoms; able to carry out all usual duties and activities
  2. Slight disability; unable to carry out all previous activities, but able to look after own affairs without assistance
  3. Moderate disability; requiring some help, but able to walk without assistance
  4. Moderately severe disability; unable to walk without assistance and unable to attend to own bodily needs without assistance
  5. Severe disability; bedridden, incontinent and requiring constant nursing care and attention
  6. Dead
Incidence of parent artery thrombosis | through 365-day post procedure
Incidence of in-construct stenosis > 50% | through 365-day post procedure
Incidence of retreatment | through 180-day and 365-day post procedure
Incidence of peri-/post-procedural serious adverse events related to the device, procedure or antiplatelet therapy | through 180-day and 365-day post procedure
Incidence of neurological death or disabling stroke | through 365-day post procedure
Incidence of complete angiographic occlusion without significant stenosis (≤ 50%), and no rebleeding or retreatment of the target aneurysm | through 365-day post procedure

CONTACTS AND LOCATIONS:
Overall Officials: David Fiorella, MD, Principal Investigator — Stony Brook University Hospital
Locations (7):
- United States (7):
  - Yale New Haven Hospital, New Haven, Connecticut
  - Wellstar Kennestone Hospital, Marietta, Georgia
  - Rush University Medical Center, Chicago, Illinois
  - University of Kentucky Albert B Chandler Hospital, Lexington, Kentucky
  - Stony Brook University Hospital, Stony Brook, New York
  - Geisinger Medical Center, Danville, Pennsylvania
  - Semmes Murphey Clinic, Memphis, Tennessee

IPD SHARING:
Plan to Share IPD: No
No individual participant data will be available.